CLINICAL TRIAL: NCT03339921
Title: Comparison of Botulinum Toxin to Fasciotomy in Treatment of Chronic Exertional Compartment Syndrome
Brief Title: Botulinum for Chronic Exertional Compartment Syndrome
Acronym: Botox
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study is being closed because it is unworkable.
Sponsor: 375th Medical Group, Scott Air Force Base (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20170037H
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Exertional Compartment Syndrome
MeSH Terms: conditions — Chronic Exertional Compartment Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum toxin injections (Experimental): Botulinum toxin injections for chronic compartment syndrome
  Interventions: Drug: Botulinum toxin injections for chronic compartment syndrome
- surgical fasciotomy (Active Comparator): surgical fasciotomy for chronic compartment syndrome
  Interventions: Procedure: surgical fasciotomy for chronic compartment syndrome

INTERVENTIONS:
Drug: Botulinum toxin injections for chronic compartment syndrome — Botulinum toxin will be injected in the upper and lower portion of the affected area with a syringe
  Arms: Botulinum toxin injections
Procedure: surgical fasciotomy for chronic compartment syndrome — linear incisions will be made into the affected compartment releasing the underlying fascial layer, reducing the pressure of the compartment
  Arms: surgical fasciotomy

SUMMARY:
We will investigate the feasibility of a simple outpatient one time injection regimen for the treatment of Chronic Exertional Compartment Syndrome (CECS). We think botulinum toxin injections will be a potentially cost-effective, low-risk alternative to surgery in reducing pain and returning patients to full activity.

DETAILED DESCRIPTION:
The study will be a prospective cohort pilot study designed to compare Active Duty patients, 18 years of age or older, with Chronic Exertional Compartment Syndrome (CECS) undergoing two different treatment interventions. The first arm will be patients receiving investigational botulinum toxin injections. The second arm will be patients who undergo the standard of care surgical fasciotomy. Both arms will be evaluated for pain relief with the universal pain scale and lower extremity functional index (LEFI) surveys at pre-treatment and again at one, three, and six months post-treatment. Clinical data that will be analyzed for research purposes in both groups include age, sex, height, weight, body mass index, time to diagnosis, minutes of exercise prior to onset of symptoms, minutes of rest before relief of symptoms, LEFI and pain on the Universal Pain Assessment Tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult ages 18-65
* Active duty military
* Unable to run 1.5 miles without producing symptoms, including aching, burning, numbness, tingling, or weakness in the affected limb
* Failed conservative treatment over a period of 2 months, including trial of rest, NSAIDs, icing, and stretching routine
* Meets standard of care clinical diagnostic intramuscular compartment pressure criteria for CECS, based on standardized IMP needle testing. See below for testing protocol and criteria.

Exclusion Criteria:

* Prior Botulinum toxin injections into the affected limb
* Prior compartment release of the affected limb
* Pregnant or becomes pregnant during the study
* Standard of care clinical exams indicating other more likely causes of leg pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Boyce, MD, Principal Investigator — Principal Investigator
Locations (1):
- 375th Medical Group, Scott Air Force Base, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Injections | Surgical Fasciotomy
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated because it is unworkable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Injections | Surgical Fasciotomy | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Functional Index
Description: The Lower Extremity Functional Index measures the functional impairment of a patient with a lower extremity disorder. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention. Score ranges from 0 to 80. Lower scores indicate more functional impairment.
Time Frame: 6 months
Population: No subjects were analyzed by a biostatistician. This study was terminated because it is unworkable. Raw data are reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Botulinum Toxin Injections | Surgical Fasciotomy
Number analyzed (Participants) | 3 | 0
score on a scale
  Lower Extremity Functional Scale Immediately Post Treatment | 57 [48 to 67] |
  Lower Extremity Functional Scale Month 1 | 60 [34 to 78] |
  Lower Extremity Functional Scale Month 2 | 62 [52 to 67] |
  Lower Extremity Functional Scale Month 6 | 55 [45 to 68] |

ADVERSE EVENTS:
Time Frame: 6 months
Description: This study was terminated because it is unworkable.
Arm/Group | Botulinum Toxin Injections | Surgical Fasciotomy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated because it is unworkable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT03339921/Prot_SAP_000.pdf